CLINICAL TRIAL: NCT06596967
Title: Home-based Heat Therapy in Older Adults with Type 2 Diabetes: a Pilot Trial
Brief Title: Heat Therapy in Type 2 Diabetes
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Bruno Roseguini, Associate Professor, Purdue University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-854; P30DK097512 (NIH)
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes
Keywords: heat therapy; type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperthermia | interventions — Diathermy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SHAM (Sham Comparator): In the sham group, water at 33ºC will be circulated through the leg sleeves.
  Interventions: Device: Sham
- HEAT THERAPY (Experimental): In the leg heat therapy group, water at 42ºC will be circulated through the leg sleeves.
  Interventions: Device: Heat therapy

INTERVENTIONS:
Device: Heat therapy — Participants will be provided with a heat therapy system comprising a controller unit with a water pump and air pump, a portable heater, and leg sleeves featuring inner-layer water-circulating pads and an outer layer of inflatable bladders. The system is engineered to facilitate effective heat transfer through gentle pneumatic inflation, accommodating various limb dimensions. The heater will be set to warm the water to 42°C. Participants will be instructed to administer the therapy for 90 minutes daily in a seated or supine position.
  Other Names: Leg heating
  Arms: HEAT THERAPY
Device: Sham — Participants will be provided with a heat therapy system comprising a controller unit with a water pump and air pump, a portable heater, and leg sleeves featuring inner-layer water-circulating pads and an outer layer of inflatable bladders. The system is engineered to facilitate effective heat transfer through gentle pneumatic inflation, accommodating various limb dimensions. The heater will warm the water to 33°C. Participants will be instructed to administer the therapy for 90 minutes daily in a seated or supine position.
  Arms: SHAM

SUMMARY:
This study aims to test whether home-based heat therapy (HT) can improve the health of older adults with type 2 diabetes (T2D). T2D is common in older adults and can lead to severe issues such as heart disease, disability, and early death. While regular exercise is known to help manage T2D, many people with the condition find it difficult to stay active. This study explores HT as a simple, non-invasive treatment that may offer similar benefits.

Participants will wear special leg sleeves that deliver heat to their legs for 90 minutes each day at home over 12 weeks. The study's primary goal is to assess whether HT treatment at home is feasible and safe to use. We hypotesize that people with diabetes who receive heat therapy will have better blood sugar control, stronger legs, less body fat, and improved ability to walk, along with lower blood pressure.

If successful, HT could offer a new option for people with T2D to manage their condition, especially for those who struggle with regular exercise. This research could lead to larger studies and help provide a practical way to improve health and quality of life for older adults with diabetes.

DETAILED DESCRIPTION:
Our objective in this proposal is to conduct a pilot randomized, sham-controlled trial to establish the feasibility, acceptability, and safety of home-based leg HT for 12 weeks in older individuals with T2D. We will also examine changes in glucose regulation, body composition, blood pressure, skeletal muscle strength, and physical function. Individuals will be asked to apply the treatment daily for 90 min using water-circulating sleeves perfused with warm water Our working hypotheses are that diabetic individuals receiving HT will manifest: 1) improved blood glucose regulation, 2) enhanced leg strength and power, 3) lower body fat content, and 4) improved walking tolerance21 and lower blood pressure.

We propose the following specific aims:

AIM 1: Establish the feasibility of home-based HT for older individuals with T2D. The primary outcomes are compliance with the HT regimen, measured by a hidden timer, completion rates, device safety, and usability.

AIM 2: Examine the effects of HT on blood glucose regulation in older adults with T2D. We will assess the change in glycated hemoglobin (HbA1c) and insulin sensitivity index (Matsuda insulin sensitivity index) between baseline and the 12-week follow-up. Glucose, insulin, and HbA1c will be measured in the Translation Core.

AIM 3: Evaluate the effect of HT on lower-extremity functioning and body composition in older adults with T2D. We will assess changes in walking endurance (6-minute walk distance), leg muscle strength and power (isokinetic dynamometry), lower extremity functioning (Short Physical Performance Battery), and body composition (Dual-energy X-ray absorptiometry).

ELIGIBILITY:
Inclusion Criteria:

1. age 55 and older
2. Type 2 Diabetes (documented by chart review, presence of treatment for type 2 Diabetes, fasting plasma glucose equal or greater than 126 mg/dL or A1C equal or greater than 6.5%).

Exclusion Criteria:

(1) HbA1c <6.5% or >9.0%, (2) body mass index > 40 kg/m2, (3) insulin-dependent Type 1 Diabetes Mellitus, (4) incident cardiovascular events in the last year (heart attack, stroke), (5) symptomatic coronary artery disease and/or heart failure, (6) uncontrolled hypertension (systolic blood pressure >150 mmHg and/or diastolic blood pressure >110 mmHg), (7) hypotension (resting systolic BP < 90 mmHg), (8) use of walking aid other than a cane, (9) active cancer, (10) impaired thermal sensation in the legs, (11) unable to fit into water-circulating garments, (12) orthopedic complications that preclude completion of physical function tests, (13) contraindications or inability to undergo a DXA scan, including implants, devices, or other foreign material, and inability to attain correct position and/or remain motionless for the measurement.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Compliance | From enrollment to the end of treatment at 12 weeks
  A built-in timer inside the pump that is inaccessible to participants will provide one assessment of patient compliance with the therapy. Compliance will be determined by dividing the number of hours of HT recorded use by the required hours. In addition, patients in both groups will receive a logbook to record their treatment sessions.
Completion rate | From enrollment to the end of treatment at 12 weeks
  Completion rates will be defined as the number of patients attending the follow-up assessments.
Safety | From enrollment to the end of treatment at 12 weeks
  The study coordinator will call patients weekly to record the occurrence of symptoms, such as faintness or dizziness after exposure to the therapy, and changes in medical status . Adverse events (AEs) will be tracked throughout the study and used as a surrogate for safety-related outcomes.

SECONDARY OUTCOMES:
Change in Insulin sensitivity | Baseline and 12-week follow-up
  Insulin sensitivity will be calculated using insulin and glucose responses during the oral glucose tolerance test
Change in blood pressure | Baseline and 12-week follow-up
  BP will be measured in triplicate in both arms using an automated monitor (Tango M2, SunTech).
Change in body composition | Baseline and 12-week follow-up
  Body composition (fat mass and fat-free mass) will be assessed via dual-energy x-ray absorptiometry (DXA).
Change in 6-minute walk distance | Baseline and 12-week follow-up
  Participants will receive standardized instructions and will be asked to walk the greatest distance possible by walking back and forth along a 100-ft corridor for 6 min.
Change in peak torque of the knee extensors | Baseline to 12-week follow-up
  Torque assessments of the knee extensors and plantar flexors will be performed using an isokinetic dynamometer (Biodex System 4 Pro, Biodex Medical Systems, Shirley, NY)
Change in Short Physical Performance Battery (SPPB) score | Baseline and 12-week follow-up
  The SPPB combines data from the usual paced 4-m walking velocity, time to rise from a seated position 5 times, and standing balance. The timed results of the subtests will be converted to an ordinal scale ranging from 0 (worst performance) to 12 (best performance).
Change in Short-Form (SF)-36 Questionnaire scores | Baseline to 12-week follow-up
  Health-related quality of life (HRQOL) will be assessed using the short-form SF-36 questionnaire, which is composed of 8 subscales.

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided